CLINICAL TRIAL: NCT01863966
Title: Efficacy and Safety Study of Hot Water Drinking Therapy in Achalasia Patients
Brief Title: Hot Water Drinking Therapy in Achalasia
Acronym: AHW
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-AchaWater
Record Dates: First submitted 2013-05-21; First posted 2013-05-29 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Achalasia
Keywords: Achalasia; Hot water drinking therapy; Pneumatic dilation
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hot water drinking therapy (Experimental): Hot water drinking before,after meal and before sleep
  Interventions: Other: hot water drinking therapy
- Pneumatic dilation (Active Comparator): Patients who are unsatisfied with hot water drinking therapy are to receive standard pneumatic dilation
  Interventions: Procedure: Pneumatic dilation

INTERVENTIONS:
Other: hot water drinking therapy — Drink 200ml hot water 3min before and after a meal. Swallow food with hot water and drink 200ml hot water before sleep
  Arms: Hot water drinking therapy
Procedure: Pneumatic dilation — Patients who are unsatisfied with hot water drinking therapy are to receive standard pneumatic dilation under endoscope
  Arms: Pneumatic dilation

SUMMARY:
From clinical observation that some achalasia patients drink water to help swallow food, the investigators have proposed a systemic hot water drinking therapy. This study is to observe its efficacy on achalasia symptoms and explore its mechanism.

DETAILED DESCRIPTION:
1. Achalasia patients will participate hot water drinking therapy: to drink 200ml of hot water before and after a meal, as well as 2 hours before sleep and to chew food carefully and swallow with hot soup.
2. Patients are followed by achalasia associated symptom scores, barium esophagram and endoscopy.
3. If patients are unsatisfied with hot water drinking therapy, they receive pneumatic dilation

ELIGIBILITY:
Inclusion Criteria:

* achalasia patients diagnosed by endoscopy, barium esophagram and manometry

Exclusion Criteria:

* could not drink water
* poor compliance
* severe comorbidities
* esophageal stenosis secondary to erosions and cancer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-03; Primary Completion 2015-11 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline achalasia symptom score at 1 month | baseline and 1 month
  Dysphagia, Regurgitation and Chest Pain scores

SECONDARY OUTCOMES:
Number of patients with adverse effects | Week 1
  adverse effects of drinking water like distention, nausea and belching
Change from baseline in barium esophagram at 1 year | baseline and 1 year
  measure esophageal diameter
Endoscopy at 1 year | year 1
  esophageal bezoars and esophageal cancer
Pneumatic dilation rate and relative efficacy | any time
  Patients who are unsatisfied with hot water drinking therapy are to receive pneumatic dilation
Change from baseline in achalasia symptom score at 1 year | baseline and 1 year
  Dysphagia,Regurgitation and Chest Pain scores
Change from baseline achalasia symptom scores at 5 years | baseline and 5 years
  Dysphagia,Regurgitation and Chest Pain scores
Change from baseline in barium esophagram at 5 years | baseline and 5 years
  measure esophageal diameter
Endoscopy at 5 years | year 5
  esophageal bezoars and esophageal cancer

CONTACTS AND LOCATIONS:
Overall Officials: Meiyun Ke, M.D., Study Director — Department of Gastroenterology, Peking Union Medical College Hospital, Chinese Academy of Medical Science
Locations (1):
- Department of Gastroenterology, Peking Union Medical College Hospital, Chinese Academy of Medical Science, Beijing, China

REFERENCES:
- [Result] Triadafilopoulos G, Tsang HP, Segall GM. Hot water swallows improve symptoms and accelerate esophageal clearance in esophageal motility disorders. J Clin Gastroenterol. 1998 Jun;26(4):239-44. doi: 10.1097/00004836-199806000-00003. PMID 9649001
- [Result] Ren Y, Ke M, Fang X, Zhu L, Sun X, Wang Z, Wang R, Wei Z, Wen P, Xin H, Chang M. Response of esophagus to high and low temperatures in patients with achalasia. J Neurogastroenterol Motil. 2012 Oct;18(4):391-8. doi: 10.5056/jnm.2012.18.4.391. Epub 2012 Oct 9. PMID 23105999